CLINICAL TRIAL: NCT03224546
Title: Cardiovascular, Immune and Psychosocial Benefits of Reduced Cocaine Use
Brief Title: Cocaine Use Reduction and Health
Acronym: RCT (04)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Randomized Clinical Trial (04); R01DA043938 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cocaine Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): This group will receive payment for providing urine samples throughout the trial.
- Low Value Alternative Reinforcer Group (Experimental): This group will receive payment for providing cocaine negative urine samples throughout the trial.
  Interventions: Behavioral: Contingency Management
- High Value Alternative Reinforcer Group (Experimental): This group will receive payment for providing cocaine negative urine samples throughout the trial.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Subjects will receive payments for providing cocaine negative urine samples.
  Arms: High Value Alternative Reinforcer Group; Low Value Alternative Reinforcer Group

SUMMARY:
Reduced drug use is a clinically meaningful target for treatment development, but few studies have evaluated the positive impacts produced by this behavioral change, preventing adoption of this endpoint in clinical trials. The proposed research will fill that critical knowledge gap by demonstrating the biopsychosocial benefits of reduced cocaine use. These data will be used to change current accepted cocaine treatment endpoints and accelerate identification of therapies for cocaine use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Self-report of recent cocaine use verified by a cocaine-positive urine sample
* Meet moderate-severe Cocaine Use Disorder Criteria
* Seeking treatment for their cocaine use
* Able to commit to 12-week intervention, plus 24-week follow up

Exclusion Criteria:

* History of serious physical or psychiatric disease (e.g., physical dependence on any drug requiring medically managed detoxification, unstable angina, uncontrolled cardiac arrhythmia, aortic stenosis, self-reported compromised immune function, extreme hypersensitivity/allergy to candida yeast or similar products, severe diagnosis for other substance use disorder) that would interfere with study participation
* Current physical or psychiatric disease that would interfere with study participation
* Poor veinous access, precluding blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Stoops, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
A formal plan for sharing final research data is not required for investigator-initiated applications with direct costs of less than $500,000. However, we felt it important to verify that the results (i.e., summary statistics and graphical/tabular representation of the data) from this study will be presented at local, regional, national and/or international conferences. In addition, a manuscript or manuscripts describing the results will be prepared for submission to a peer-reviewed journal or journals, and the final, accepted version(s) of the manuscript(s) will be submitted to PubMed Central. As requested, the final research data will be made available to oversight or regulatory committees. The rights and privacy of individuals who participated will be protected at all times, and at no time will identifiers be included that would permit linkages to the individual subjects and variables that could lead to deductive disclosure of the identity of subjects.

REFERENCES:
- [Derived] Ferretti ML, Regnier SD, Irons JG, Stoops WW. Polysubstance use patterns and risk behaviors among people with cocaine use disorder. Exp Clin Psychopharmacol. 2025 Dec;33(6):586-593. doi: 10.1037/pha0000813. PMID 41343351
- [Derived] Stoops WW, Shellenberg TP, Regnier SD, Cox DH, Adatorwovor R, Hays LR, Anderson DM, Lile JA, Schmitz JM, Havens JR, Segerstrom SC. Influence of cocaine use reduction on markers of immune function. J Neuroimmunol. 2024 Dec 15;397:578470. doi: 10.1016/j.jneuroim.2024.578470. Epub 2024 Oct 28. PMID 39504756
- [Derived] Regnier SD, Shellenberg TP, Koffarnus MN, Cox DH, Lile JA, Rush CR, Stoops WW. Cocaine abstinence during the "critical period" of a contingency management trial predicts future abstinence in people with cocaine use disorder. Drug Alcohol Depend. 2023 Dec 1;253:111030. doi: 10.1016/j.drugalcdep.2023.111030. Epub 2023 Nov 18. PMID 38006674

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Started | 42 | 41 | 44
Completed | 26 | 19 | 29
Not Completed | 16 | 22 | 15
Not completed — Lost to Follow-up | 9 | 8 | 3
Not completed — Withdrawal by Subject | 7 | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group | Total
Number analyzed (Participants) | 42 | 41 | 44 | 127
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 44 | 127
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 15 | 43
  Male | 29 | 26 | 29 | 84
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 32 | 34 | 34 | 100
  White | 10 | 5 | 5 | 20
  More than one race | 0 | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 44 | 127

OUTCOME MEASURES:

1. Primary Outcome: Endothelin-1 Levels
Description: Endothelin-1 levels will be measured. They will be recorded in pg/ml.
Time Frame: At baseline.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 42 | 41 | 44
pg/ml | 2.15 (.784) | 2.063 (.699) | 1.956 (.606)

2. Primary Outcome: Endothelin-1 Levels
Description: Endothelin-1 levels will be measured. They will be recorded in pg/ml.
Time Frame: Week 6 of study participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 23 | 16 | 29
pg/ml | 1.886 (.759) | 1.923 (.478) | 1.939 (.718)

3. Primary Outcome: Endothelin-1 Levels
Description: Endothelin-1 levels will be measured. They will be recorded in pg/ml.
Time Frame: Week 12 of study participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 16 | 26
pg/ml | 2.093 (0.673) | 2.083 (.772) | 2.086 (.680)

4. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure is recorded during participant visits and is recorded in mm Hg
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 42 | 41 | 44
mm Hg | 96.69 (15.77) | 97.22 (12.94) | 97.08 (11.93)

5. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 1 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 34 | 31 | 34
mm Hg | 99.22 (16.45) | 99.66 (13.24) | 97.38 (13.18)

6. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 2 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 31 | 27 | 33
mm Hg | 95.92 (15.85) | 99.78 (9.85) | 97.07 (14.03)

7. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 3 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 29 | 25 | 36
mm Hg | 97 (13.57) | 100.5 (12.39) | 96.18 (12.06)

8. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 4 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 27 | 24 | 27
mm Hg | 97.28 (15.08) | 102.02 (12.99) | 98.66 (12.41)

9. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 5 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 27 | 25 | 31
mm Hg | 96.12 (14.78) | 99.72 (14.33) | 97.96 (13.18)

10. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 6 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 27 | 25 | 31
mm Hg | 97.46 (13.51) | 100.93 (11.70) | 95.40 (13.23)

11. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 7 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 25 | 21 | 28
mm Hg | 94.72 (14.88) | 100.13 (11.28) | 92.59 (12.29)

12. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 8 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 26 | 21 | 26
mm Hg | 96.14 (14.84) | 100.05 (14.46) | 94.55 (12.38)

13. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 9 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 24 | 17 | 29
mm Hg | 100.02 (16.59) | 100.19 (10.81) | 94.46 (12.21)

14. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 10 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 29 | 16 | 25
mm Hg | 99.43 (17.18) | 102.68 (11.80) | 95.71 (13.60)

15. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 11 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 20 | 19 | 26
mm Hg | 98.06 (15.53) | 101.31 (12.07) | 93.20 (11.05)

16. Primary Outcome: Mean Arterial Pressure
Description: Mean Arterial Pressure was recorded during subject visits and is recorded in mm Hg
Time Frame: Week 12 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 23 | 18 | 26
mm Hg | 97.98 (14.21) | 102.10 (11.00) | 93.05 (11.89)

17. Secondary Outcome: Interleukin-10
Description: Interleukin-10 levels will be measured throughout subject participation. They will be recorded in pg/ml.
Time Frame: At baseline.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 42 | 41 | 44
pg/ml | .547 (.750) | .429 (.424) | .251 (.106)

18. Secondary Outcome: Interleukin-10
Description: Interleukin-10 levels will be measured throughout subject participation. They will be recorded in pg/ml.
Time Frame: Week 6 of study participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 23 | 16 | 29
pg/ml | .587 (1.23) | .329 (.116) | .257 (.102)

19. Secondary Outcome: Interleukin-10
Description: Interleukin-10 levels will be measured throughout subject participation. They will be recorded in pg/ml.
Time Frame: Week 12 of study participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 16 | 26
pg/ml | .384 (.663) | .481 (.514) | .230 (.907)

20. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 42 | 41 | 44
minutes | 393.81 (135.91) | 379.27 (139.21) | 353.18 (118.31)

21. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 1 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 34 | 31 | 41
minutes | 397.53 (135.60) | 413.45 (112.50) | 393.16 (121.13)

22. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 2 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 31 | 27 | 33
minutes | 420.74 (149.37) | 447.76 (141.53) | 388.14 (136.68)

23. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 3 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 29 | 25 | 36
minutes | 424.45 (145.55) | 414.5 (144.60) | 393.78 (110.19)

24. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 4 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 27 | 24 | 27
minutes | 415.22 (149.02) | 390.10 (149.14) | 360.37 (132.39)

25. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 5 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 27 | 25 | 31
minutes | 430.23 (119.61) | 426.49 (157.00) | 360 (144.31)

26. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 6 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 26 | 21 | 32
minutes | 444.08 (108.42) | 394.46 (143.41) | 379.94 (120.34)

27. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 7 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 25 | 21 | 28
minutes | 437.57 (99.48) | 421.11 (190.85) | 384.78 (118.26)

28. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 8 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 26 | 21 | 26
minutes | 452.89 (117.21) | 395.74 (171.67) | 386.29 (130.64)

29. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 9 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 24 | 17 | 30
minutes | 458.13 (123.29) | 426.67 (144.25) | 387.69 (135.79)

30. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 10 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 25 | 16 | 29
minutes | 453.28 (95.52) | 405.44 (160.29) | 373.21 (148.41)

31. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 11 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 20 | 19 | 26
minutes | 441.51 (96.25) | 389.79 (185.49) | 370.16 (144.97)

32. Secondary Outcome: Total Sleep Time
Description: Sleep time the night before in minutes
Time Frame: Week 12 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 23 | 18 | 26
minutes | 435 (136.74) | 378.23 (150.62) | 387.05 (137.55)

33. Secondary Outcome: Hamilton Depression Scale Score
Description: Score on the Hamilton Depression Inventory. Higher scores indicate greater depression symptoms. Minimum = 0, Maximum =56.
Time Frame: At baseline
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 42 | 41 | 44
score on a scale | 4 [0 to 10] | 3 [0 to 7] | 5.5 [0 to 12.75]

34. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 1 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 30 | 22 | 33
score on a scale | 2 [0 to 6] | 1.5 [0 to 6.5] | 4 [0 to 9]

35. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 2 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 24 | 19 | 27
score on a scale | 1 [0 to 4] | 2 [0 to 5.5] | 3 [0 to 10]

36. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 3 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 26 | 20 | 25
score on a scale | 1 [0 to 4.75] | 1 [0 to 4] | 3 [0 to 8]

37. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 4 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 17 | 24
score on a scale | 1 [0 to 4] | 1 [0 to 5] | 2.5 [0 to 6.75]

38. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 5 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 24 | 19 | 28
score on a scale | 1 [0 to 4] | 1 [0 to 4] | 2 [0 to 6]

39. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 6 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 23 | 17 | 29
score on a scale | 0 [0 to 2.5] | 1 [0 to 4] | 1 [0 to 5]

40. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 7 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 22 | 16 | 21
score on a scale | 1 [0 to 4.75] | 1.5 [0 to 4.75] | 0 [0 to 2]

41. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 8 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 18 | 21
score on a scale | 2 [0 to 6] | 1 [0 to 2.75] | 1 [0 to 5]

42. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 9 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 15 | 22
score on a scale | 1 [0 to 4] | 0 [0 to 2.5] | 0.5 [0 to 2.25]

43. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 10 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 19 | 15 | 23
score on a scale | 1 [0 to 8.5] | 0 [0 to 1.5] | 1 [0 to 6]

44. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 11 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 19 | 18 | 20
score on a scale | 1 [0 to 4] | 0 [0 to 2.75] | 1 [0 to 7]

45. Secondary Outcome: Hamilton Depression Scale Score
Description: as for outcome 33
Time Frame: Week 12 of Participation
Population: Available participants to be measured.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 17 | 26
score on a scale | 1 [0 to 3] | 0 [0 to 1] | 0 [0 to 3.75]

46. Secondary Outcome: Criteria for Cocaine Use Disorder Diagnosis
Description: Number of criteria met on a Structured Clinical Interview as endorsed yes/no on a series of 11 questions on a scale. Range = 0-11. Higher scores indicate greater severity of Cocaine Use Disorder (e.g., more life problems due to cocaine use).
Time Frame: At Baseline
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: number of criteria met
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 42 | 41 | 44
number of criteria met | 8.4 (1.9) | 7.2 (2.0) | 8.6 (1.8)

47. Secondary Outcome: Criteria for Cocaine Use Disorder Diagnosis
Description: as for outcome 46
Time Frame: Week 12 of Participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: number of criteria met
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 21 | 17 | 26
number of criteria met | 6.2 (3.2) | 4.8 (2.7) | 6.5 (2.2)

48. Secondary Outcome: Reactive Hyperemia Index
Description: Measure of peripheral arterial tonomotry which assesses peripheral microvascular function through changes in amplitude of pulses in fingertips. Reactive hyperemia index (RHI) is "determined by calculating the ratio of hyperemic pressure (RHm) to baseline pressure (BLm) in the measurement and control arms (RHc and BLc respectively)" (Rosenberry and Nelson, 2020). This yields a natural log RHI ratio with higher scores indicating worse microvascular function. Being calculated as a natural log, there range is infinite.
Time Frame: At Baseline
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: ln(ratio)
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 38 | 37 | 38
ln(ratio) | .61 (.32) | .63 (.33) | .51 (.41)

49. Secondary Outcome: Reactive Hyperemia Index
Description: Measure of peripheral arterial tonomotry which assesses peripheral microvascular function through changes in amplitude of pulses in fingertips. Reactive hyperemia index (RHI) is "determined by calculating the ratio of hyperemic pressure (RHm) to baseline pressure (BLm) in the measurement and control arms (RHc and BLc respectively)" (Rosenberry and Nelson, 2020). This yields a natural log RHI ratio with higher scores indicating worse microvascular function. This yields a natural log RHI ratio with higher scores indicating worse microvascular function. Being calculated as a natural log, there range is infinite.
Time Frame: Week 12 of participation
Population: Available participants to be measured.
Measure: Mean (Standard Deviation); unit: ln(ratio)
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
Number analyzed (Participants) | 20 | 17 | 23
ln(ratio) | .53 (.37) | .81 (.40) | .42 (.54)

ADVERSE EVENTS:
Time Frame: 12 week clinical trial participation
Arm/Group | Control Group | Low Value Alternative Reinforcer Group | High Value Alternative Reinforcer Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 17/42 | 15/41 | 20/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=42) | Low Value Alternative Reinforcer Group (N=41) | High Value Alternative Reinforcer Group (N=44)
Abnormal ECG (Cardiac disorders) | 8 (8) | 8 (8) | 10 (10)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Elevated Creatine Kinase (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Difficult Blood Draw (Vascular disorders) | 3 (3) | 1 (1) | 3 (3)
Unusual/Unpleasant Skin Sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03224546/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT03224546/ICF_000.pdf